CLINICAL TRIAL: NCT07296250
Title: A Randomized, Prospective Phase II Clinical Trial - Extended Chemotherapy or Not Based on Circulating Tumor Cell Counts in Postoperative ENE-Positive Oral Cavity Cancer Patients After Completing Adjuvant Concurrent Chemoradiotherapy
Brief Title: Circulating Tumor Cell Counts in Postoperative ENE-Positive Oral Cavity Cancer Patients After Adjuvant CCRT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chun-Ta Liao, Professor Attending Physicians, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 202402125B0
Record Dates: First submitted 2025-11-21; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Head and Neck Cancer; Oral Cancer
Keywords: oral cancer; ENE; Circulating tumor cells; Adjuvant concurrent Chemoradiation, adjuvant CCRT; Circulating tumor microemboli (CTM)
MeSH Terms: conditions — Head and Neck Neoplasms; Mouth Neoplasms; Neoplastic Cells, Circulating | interventions — Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention): participants without low-dose oral chemotherapy. Each patient must continue to be tracked for ENE or other postoperative risks for one year, and with blood testing every tree month.
- experimental (Experimental): participants with low-dose oral chemotherapy. Each patient must continue to be tracked for ENE or other postoperative risks for one year, and with blood testing every tree month.
  Interventions: Procedure: low-dose oral chemotherapy

INTERVENTIONS:
Procedure: low-dose oral chemotherapy — recruit 100 oral cavity cancer patients with ENE or other postoperative risks.10 mL of research blood was drawn four times in total.Each patient must continue to be tracked for ENE or other postoperative risks for one year, and with blood testing every tree month.
  Arms: experimental

SUMMARY:
The aim 1 of this trial is the development of the Circulating tumor cells (CTCs) definition of oral cancer minimal residual disease (MRD), and aim 2 is a prospective trial of oral cancer treatment. If this trial is successful, it is expected that it may be able to provide a standard diagnostic tool (MRD in Oral Cavity Squamous Cell Carcinoma (OCSCC)) and treatment mode (extended adjuvant chemotherapy with low-dose oral chemotherapy). The survival rate of patients will be improved.

DETAILED DESCRIPTION:
The aim 1 of this trial is the development of the CTC definition of oral cancer MRD, and aim 2 is a prospective trial of oral cancer treatment. If this trial is successful, it is expected that it may be able to provide a standard diagnostic tool (MRD in OCSCC) and treatment mode (extended adjuvant chemotherapy with low-dose oral chemotherapy). The survival rate of patients will be improved.

This three-year study is expected to recruit 100 oral cavity cancer patients with extracapsular nodal extension (ENE) or other postoperative risks.10 mL of research blood was drawn four times in total.Each patient must continue to be tracked for ENE or other postoperative risks for one year, and with blood testing every tree month.

For the negative selection of CTCs by the negative selection system. For the positive selection of CTCs by counting Epithelial cell adhesion molecule(EpCAM)-positive and Hoechst-positive cells under a microscope with a hemocytometer.

In brief, CTC could predict a poor prognosis in HNSCC patients. But the role of longitudinal CTC follow-up in ENE+ oral cavity cancer patients remains unclear.

ELIGIBILITY:
Inclusion Criteria:

Participants with Cancer:

1. Aged between 18 and 90 years.
2. Histologically confirmed diagnosis of head and neck squamous cell carcinoma (HNSCC).
3. Completed surgical treatment and identified as having high-risk factors, followed by concurrent chemoradiotherapy.
4. Willing to continue follow-up visits at the hospital after completion of treatment.

Exclusion Criteria:

1. Presence of psychiatric disorders.
2. Deemed unsuitable for participation by the attending physician.
3. Unwilling to participate in the study.

Ages: 18 Months to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Circulating tumor cells (CTCs) testing | baseline
  participants will undergo CTCs testing after completing concurrent Chemoradiotherapy (CCRT). If CTC-positive (≥5.0 cells/mL), participants will receive low-dose oral chemotherapy for three months, followed by repeat CTC testing. Persistent positivity will warrant continued treatment up to one year after curative surgery, while negativity will lead to treatment discontinuation.
Circulating tumor cells (CTCs) testing | 3 month
  participants will undergo CTCs testing after completing concurrent Chemoradiotherapy (CCRT). If CTC-positive (≥5.0 cells/mL), participants will receive low-dose oral chemotherapy for three months, followed by repeat CTC testing. Persistent positivity will warrant continued treatment up to one year after curative surgery, while negativity will lead to treatment discontinuation.
Circulating tumor cells (CTCs) testing | 6 month
  participants will undergo CTCs testing after completing concurrent Chemoradiotherapy (CCRT). If CTC-positive (≥5.0 cells/mL), participants will receive low-dose oral chemotherapy for three months, followed by repeat CTC testing. Persistent positivity will warrant continued treatment up to one year after curative surgery, while negativity will lead to treatment discontinuation.
Circulating tumor cells (CTCs) testing | 9 month
  participants will undergo CTCs testing after completing concurrent Chemoradiotherapy (CCRT). If CTC-positive (≥5.0 cells/mL), participants will receive low-dose oral chemotherapy for three months, followed by repeat CTC testing. Persistent positivity will warrant continued treatment up to one year after curative surgery, while negativity will lead to treatment discontinuation.

CONTACTS AND LOCATIONS:
Overall Officials: ChunTa Liao, PhD, Principal Investigator — Division of Otolaryngology, Chang Gung Memorial Hospital
Locations (1):
- Linkou Chang Gung Memorial Hospital, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided